CLINICAL TRIAL: NCT04538092
Title: Single Institution Prospective Analysis of an Enhanced Recovery After Complex Spine Surgery Protocol
Brief Title: Complex Spine Enhanced Recovery After Surgery (ERAS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moved to different institution
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Spine Society (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-1705
Record Dates: First submitted 2020-08-20; First posted 2020-09-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-10

CONDITIONS: Scoliosis Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard post op complex spine orders placed for patients undergoing deformity correction
- ERAS (Experimental): Enhanced recovery after surgery protocol is applied to the patients undergoing deformity correction
  Interventions: Other: Enhanced Recovery After Surgery Protocol

INTERVENTIONS:
Other: Enhanced Recovery After Surgery Protocol — The investigators have developed an Enhanced Recovery After Surgery protocol for complex spine surgery at UNC. This study will help elucidate the effects of multiple interventions tailored to help patients recover from complex surgery.
  Other Names: Preoperative education; Preoperative nutrition; Intraoperative analgesia; Intraoperative fluid resuscitation; Postoperative analgesic; Postoperative mobilization; Postoperative nutrition; Preoperative screening; Postoperative antibiotics; Preoperative analgesia
  Arms: ERAS

SUMMARY:
In the field of Adult Spinal Deformity (ASD), there are currently no standardized protocols for preoperative, intraoperative or post-operative care. New standards are being created for minimally invasive spine surgery within orthopedics and some neurosurgical centers. This study will evaluate the efficacy of an Enhanced Recovery After Surgery protocol for complex spine surgery performed for the treatment of ASD.

DETAILED DESCRIPTION:
Purpose : In the field of Adult Spinal Deformity (ASD), there are currently no standardized protocols for preoperative, intraoperative or post-operative care. New standards are being created for minimally invasive spine surgery within orthopedics and some neurosurgical centers. This study will evaluate the efficacy of an Enhanced Recovery After Surgery protocol for complex spine surgery performed for the treatment of ASD.

Participants : Patients undergoing surgery aimed at treating adult spinal deformity are the subject of this research. This population was chosen as these procedures are often associated with prolonged length of stay (LOS), high post-operative narcotic use, and often require complex post-operative discharge planning.

Procedures : Patients undergoing surgery to address the complications of ASD present a unique challenge in that this patient population is diverse, and there are multiple operative procedures available to treat the same condition. Given that there are currently no accepted or recommended Enhanced Recovery After Surgery protocols for complex spine procedures, the investigators have developed an ERAS protocol at the University of North Carolina (UNC) in collaboration with the anesthesia department for the support of complex surgical patients.

Hypothesis: Implementing a multi-modal enhanced recovery after complex spine surgery protocol will improve patient measured outcomes and patient functional outcomes leading to a statistically significant reduction in LOS, post-operative pain, complication rate, cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of the International Statistical Classification of Diseases and Related Health Problems (ICD-10) Scoliosis (M41.9) category.
* Patients undergoing a > 5 level arthrodesis using one of the following Current Procedural Terminology (CPT) coded procedures 22534, 22585, 22614, 22632, 22634 with either 22842, 22853
* Cobb angle > 10 degrees
* Failure of 3 months of conservative management

Exclusion Criteria:

* Prior scoliosis surgery not performed at UNC Chapel Hill Hospital Facilities
* Deformity correction due to trauma
* History of neoplastic spine disease
* Patients with active osteomyelitis
* Patients with prior cement augmentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Length of Stay | From conclusion of surgery to hospital discharge, an expected average of 10 days
  Number of nights spent in the hospital following surgery

SECONDARY OUTCOMES:
Narcotic usage | From conclusion of surgery to 12 months
  Total morphine milligram equivalents (MME) utilized while inpatient and after discharge
30 Day Readmission | From day of hospital discharge to 30 days
  Did the patient require a repeat hospitalization within 30 days after the initial surgery?
90 Day Readmissions | From day of hospital discharge to 90 days
  Did the patient require a repeat hospitalization within 90 days after the initial surgery
30 Day Reoperations | From day of hospital discharge to 30 days
  Did the patient require a repeat reoperation within 30 days after the initial surgery
Change in Oswestry Disability Index Score from Pre-op baseline. | Preop to post op comparison of ODI at 4 days, 2 weeks, 6 weeks, 12 weeks and 6 months.
  The Oswestry Disability Index (ODI) for functional impairment is used to quantify disability related to lower back pain. The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound. Higher scores reflect more severe disability.
  The Oswestry Disability Index (ODI) measures patients' degree of disability related to lower back pain. The ODI has 10 items (Pain, self-care, bring, walking, sitting, standing, sleeping, sex, social, and travelling). After adding up the total score of each item, the initial total score is 0 to 50 points. Then divide the total score by 5 and multiply by 20 to get the final score of 0 to 100.
Promis Score - Pain | Preop to post op comparison of PROMIS instruments at 6 weeks and 6 months.
  Patient-Reported Outcomes Measurement Information System (PROMIS), this 8-item, self-reported tool will assess a person's level of confidence to manage/control symptoms, to manage their symptoms in different settings and to keep symptoms from interfering with work, sleep, relationships or recreational activities. Each question usually has five response options ranging in value from 1 to 5. The total raw score for a measure is converted to into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. A higher PROMIS T-score represents more of the concept being measured.
Promis Score - Physical Activity | Preop to post op comparison of PROMIS instruments at 6 weeks and 6 months.
  Patient-Reported Outcomes Measurement Information System (PROMIS), this 8-item, self-reported tool will assess a person's level of confidence to manage/control symptoms, to manage their symptoms in different settings and to keep symptoms from interfering with work, sleep, relationships or recreational activities. Each question usually has five response options ranging in value from 1 to 5. The total raw score for a measure is converted to into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. A higher PROMIS T-score represents more of the concept being measured.
Promis Score - Physical Function | Preop to post op comparison of PROMIS instruments at 6 weeks and 6 months.
  Patient-Reported Outcomes Measurement Information System (PROMIS), this 8-item, self-reported tool will assess a person's level of confidence to manage/control symptoms, to manage their symptoms in different settings and to keep symptoms from interfering with work, sleep, relationships or recreational activities. Each question usually has five response options ranging in value from 1 to 5. The total raw score for a measure is converted to into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. A higher PROMIS T-score represents more of the concept being measured.
Time to mobilization | From the end of surgery until the date of hospital discharge, assessed up to 1 month.
  The amount of time needed from the completion of surgery until the patient is ambulating out of bed
Time to oral intake | From the end of surgery until the date of oral intake, assessed up to 2 weeks.
  The amount of time needed from the completion of surgery until the patient is able to take food or drink orally
Change in Coronal Cobb Angle | Within 6 months pre-operatively and up to 6 months postoperatively
  Standard radiographic description of standing scoliosis x-ray made using the Cobb angle measured in degrees. Assessed pre and post-operatively at 2, 6, and 12 weeks and 6 months
Change in Degrees of Apical Vertebra Rotation | Within 6 months pre-operatively and up to 6 months postoperatively
  Standard radiographic description of the change between standing scoliosis x-ray made using the Apical Vertebra's Rotation measured in degrees. Assessed pre and post-operatively at 2, 6, and 12 weeks and 6 months
Change in Thoracic Kyphosis (TK) | Within 6 months pre-operatively and up to 6 months postoperatively
  Standard radiographic description of standing scoliosis x-ray made using the Thoracic Kyphosis (TK) measured in degrees. Assessed pre and post-operatively at 2, 6, and 12 weeks and 6 months
Change in Lumbar Lordosis (LL) | Within 6 months pre-operatively and up to 6 months postoperatively
  Standard radiographic description of standing scoliosis x-ray made using the Lumbar Lordosis (LL) measured in degrees. Assessed pre and post-operatively at 2, 6, and 12 weeks and 6 months
Change in Sacral Slope (SS) | Within 6 months pre-operatively and up to 6 months postoperatively
  Standard radiographic description of standing scoliosis x-ray made using the Sacral Slope (SS) measured in degrees. Assessed pre and post-operatively at 2, 6, and 12 weeks and 6 months
Change in Pelvic Tilt (PT) | Within 6 months pre-operatively and up to 6 months postoperatively
  Standard radiographic description of standing scoliosis x-ray made using the Pelvic Tilt (PT) measured in degrees. Assessed pre and post-operatively at 2, 6, and 12 weeks and 6 months
Change in Pelvic Incidence (PI) | Within 6 months pre-operatively and up to 6 months postoperatively
  Standard radiographic description of standing scoliosis x-ray made using the Pelvic Incidence (PI) measured in degrees. Assessed pre and post-operatively at 2, 6, and 12 weeks and 6 months
Change in Sagittal Vertical Axis (SVA) Measurement | Within 6 months pre-operatively and up to 6 months postoperatively
  Sagittal Vertical Axis (SVA) measurement assessed using standing scoliosis x-ray and reported in centimeters
Change in Coronal Imbalance Measurement | Within 6 months pre-operatively and up to 6 months postoperatively
  Coronal Imbalance measurement assessed using standing scoliosis x-ray and reported in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Abumoussa, MD MSc, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Deidentified individual data that supports the results will be shared beginning 36 months following publication
Access Criteria: An investigator who proposes to use the data must have approval from an IRB, IEC, or REB, as applicable and an executed data use/sharing agreement with UNC.